CLINICAL TRIAL: NCT05326763
Title: Functional and Electromyographical Changes After Platelet Rich Plasma or Dextrose Injection in Chronic Lateral Epicondylitis
Brief Title: Functional and Electromyographical Changes After PRP or Dextrose Injection in Chronic Lateral Epicondylitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chen Yueh (Other)
Responsible Party: Sponsor-Investigator, Chen Yueh, Principal Investigator, Sin-Lau Hospital
Organization: Sin-Lau Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLH-M109-01
Record Dates: First submitted 2021-09-13; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Tennis Elbow
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- platelet rich plasma group (Active Comparator): Preparing 2 mL of PRP with concentration of 4-6 times the average normal values, 20mL of blood will be first collected from the patient's upper limb cubital vein using an 18G needle.
  Interventions: Drug: Platelet Rich Plasma
- dextrose group (Active Comparator): 4 ml of PRP + 4 ml of 0.9% saline -h 2 ml of 1% lidocaine (10-ml syringe).
  Interventions: Drug: Dextrose 50%
- Placebo (the control group) (No Intervention)

INTERVENTIONS:
Drug: Platelet Rich Plasma — Preparing 2 mL of PRP with concentration of 4-6 times the average normal values, 20mL of blood will be first collected from the patient's upper limb cubital vein using an 18G needle. A local subcutaneous anesthesia (2 ml of 1% lidocaine) will be finished by the orthopedist.
  Arms: platelet rich plasma group
Drug: Dextrose 50% — The group will use 4 ml of PRP + 4 ml of 0.9% saline -h 2 ml of 1% lidocaine (10-ml syringe).
  Arms: dextrose group

SUMMARY:
The purpose of this study is to find out functional and electromyographical changes after platelet rich plasma and dextrose injection in chronic lateral epicondylitis.

DETAILED DESCRIPTION:
Both platelet rich plasma (PRP) and dextrose treat chronic lateral epicondylalgia (CLE), mechanically by enhancing tendon cell proliferation, differentiation, and maturation. In fact, hypertonic glucose injection is much cost-effective as compared to PRP. Hence, it is of clinical value to compare the recovery of extensor carpi radialis breveis (ECRB) muscular structure and muscular function between PRP and hypertonic glucose injection.

The investigators will measure functional outcome and force gradation after PRP and glucose injection in CLE patients using multi-electromyography, functional score (Disabilities of the Arm, Shoulder and Hand (DASH) and Patient-Rated Tennis Elbow Evaluation (PRTEE)) and force (gripping power and maximal voluntary contraction (MVC) during wrist extension) before and 12 weeks after injection. The hypotheses of this study are 1) lower MVC and greater force fluctuations of a force task in the affected muscle in individuals with CLE; 2) lower discharge rate and higher discharge variability of motor units of a force task in the affected muscle in individuals with CLE than those in the contralateral sound side; 3) the PRP group shows a greater improvement in a visual analog scale (VAS), DASH, PRTEE score, MVC, and the size of force fluctuations than the glucose group after treatment. 4) the PRP group shows a greater discharge rate and lower discharge variability for a force task than the glucose group after treatment.

ELIGIBILITY:
The control group

Inclusion criteria:

1. The ages of 20-65 years without any neurological or muscular disease.

Exclusion criteria:

1. Systemic disorders such as diabetes, rheumatoid arthritis, or hepatitis

The treatment group (Experimental group)

Inclusion Criteria:

1. Patients with lateral epicondylitis in the elbow (age: 20-65 years old)
2. Pain unresponsive to 1 of 3 conventional therapy programs (local steroid injections, physical/occupational therapy, nonsteroidal anti-inflammatory medications)
3. History of elbow pain for at least 3 months
4. Elbow pain at least 50 mm/100 mm using a visual analog scale (VAS)

Exclusion Criteria:

1. Healthy population between the ages of 20-65 years
2. Pregnancy
3. History of bleeding disorder, anemia, or any blood disorder (such as Hemoglobin <11 g/dL; Hematocrit <33%; Platelet count outside of the normal range of 150 to 400 x1000/u)
4. Active bilateral elbow tendinosis within 4 weeks, previous surgery for elbow tendinosis or fracture of the affected elbow
5. History of arthritis or, cervical radiculopathy, carpal tunnel syndrome on the affected side within 1 year before randomization
6. Systemic disorders such as diabetes, rheumatoid arthritis, or hepatitis
7. Uncooperative patient or patient with neurological disorders who is incapable of following directions or who is predictably unwilling to return for follow-up examinations
8. Hypothyroidism
9. Received local steroid injections within 6 weeks, physical/occupational therapy within 4 weeks, or non- steroidal anti-inflammatory medications within 1 week
10. Intolerance to acetaminophen

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score on a visual analog scale (VAS) | 12 weeks
  a 10 cm line with anchor statements on the left (no pain) and on the right (extreme pain)
Disabilities of the Arm, Shoulder and Hand (DASH) score | 12 weeks
  scored 0 (no disability) to 100
Patient-Rated Tennis Elbow Evaluation (PRTEE) score | 12 weeks
  pain and disability from 0 to 10(0 = no difficulty, 10 = unable to do)
Level of force | 12 weeks
  extension of maximal voluntary contraction
Level of force | 12 weeks
  gripping power
The gradation of muscle force(the surface electromyogram) | 12 weeks
  the number of motor units active

CONTACTS AND LOCATIONS:
Overall Officials: Yueh Chen, Principal Investigator — Madou Sin-Lau Hosptial, the Presbyterian Church in Taiwan
Locations (1):
- Chen Yueh, Tainan, Taiwan